CLINICAL TRIAL: NCT00000422
Title: Subgroups of FMS: Symptoms, Beliefs and Tailored Treatments
Brief Title: Tailored Treatments of Fibromyalgia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Dennis Turk, Study Principal Investigator, University of Washington
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 14866-D; R01AR044724 (NIH); NIAMS-036
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2013-10-30 (Estimated); Status verified 2013-10

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia Syndrome (FMS); Physical therapy; Psychotherapy; Group counseling; Human therapy relations; Interpersonal relations; Chronic pain; Cognition; Emotion; Memory; Musculoskeletal disorder; Psychological stressor; Psychological adaptation; Outcomes research
MeSH Terms: conditions — Fibromyalgia; Chronic Pain; Musculoskeletal Diseases; Stress, Psychological | interventions — Exercise

INTERVENTIONS:
Behavioral: Cognitive-behavioral psychotherapy and physical exercise

SUMMARY:
This study will evaluate the effects of matching treatments to people with fibromyalgia syndrome (FMS) on the basis of their psychosocial and behavioral characteristics. We will look at how patients respond to a rehabilitation program that includes physical therapy and information about fibromyalgia. We will combine this program with psychological treatments that are either matched or mismatched to the way patients cope with and adapt to symptoms of FMS. The second aim of our study is to better understand how different FMS symptoms may vary together and how these symptoms change as a result of treatment in a person's natural environment. People with FMS and healthy people of the same ages will record their moods, thoughts, symptoms, activities, and fatigue levels three times a day for 2 weeks. Participants will use palm-top computers to record these "real-time" assessments. This approach will permit people to rate how they feel at a particular time rather than looking back in time.

DETAILED DESCRIPTION:
Fibromyalgia syndrome (FMS) is a prevalent, chronic musculoskeletal pain disorder. Despite extensive study, researchers do not understand well the etiology and pathophysiologic mechanisms of FMS, and have not shown any treatment to be universally effective. We propose that FMS is a complex disorder involving multiple factors, both physical and psychosocial-behavioral.

In our previous research, we demonstrated that FMS patients are heterogeneous in the psychosocial-behavioral axis and can be classified into three distinct subgroups on the basis of their psychosocial adaptation to symptoms. In this study we will extend our previous research and attempt to match treatments to patients' psychosocial-behavioral characteristics. Specifically, we will test the efficacy of uniquely tailored treatment for each psychosocial subgroup.

We will treat three groups of FMS patients with one of three treatment protocols involving standard physical therapy and varying psychological treatments. A total of 312 FMS patients will undergo six half-day interdisciplinary treatment sessions consisting of psychological treatments and physical therapy emphasizing aerobic conditioning, pacing, and body mechanics. All protocols include a standardized physical therapy and either cognitive-behavioral pain management therapy, interpersonal skill training, or supportive counseling.

In addition to the treatment outcome study, we will prospectively assess various symptoms of FMS in the patients' natural habitats to better understand covariations of FMS symptoms. Patients will do repeated daily monitoring using a palm-top computer (ecological momentary assessment), which will permit us to evaluate process ratings compared to retrospective reports.

Overall, the results of these studies should establish the benefit of matching treatments to patient characteristics and enhance our understanding of the roles of cognitive-affective-behavioral adaptation by people with FMS.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Able to visit Seattle based clinic 9 times
* Meet ACR criteria for FMS

Exclusion Criteria:

* Pregnancy
* Exercise contraindicated by physician due to other medical conditions
* Significant psychopathology
* Do not meet FMS criteria
* Cardiac problems

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312
Dates: Start 1998-07; Primary Completion 2004-05 (Actual); Study Completion 2004-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis C. Turk, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- [Result] Burwinkle T, Robinson JP, Turk DC. Fear of movement: factor structure of the tampa scale of kinesiophobia in patients with fibromyalgia syndrome. J Pain. 2005 Jun;6(6):384-91. doi: 10.1016/j.jpain.2005.01.355. PMID 15943960
- [Result] Robinson JP, Turk DC. Relations between self-reports and physical performance among fibromyalgia syndrome patients. J Pain 4, Number 2 (Suppl 1): 15, 2002.
- [Result] Turk DC, Robinson JP. Predictors of self-reported activity level and activity limitations in fibromyalgia syndrome. J Pain 4, Number 2 (Suppl 1): 16, 2003.
- [Result] Turk DC, Robinson JP, Burwinkle T. Prevalence of fear of pain and activity in patients with fibromyalgia syndrome. J Pain. 2004 Nov;5(9):483-90. doi: 10.1016/j.jpain.2004.08.002. PMID 15556826
- [Result] Burwinkle T, Robinson JP, Turk DC. The role of physical, demographic, and psychological factors in symptom reporting and treatments of fibromyalgia syndrome patients. J Pain 6 (Suppl 1), S79, 2005.